CLINICAL TRIAL: NCT06750250
Title: The Effects of Aerobic Exercise on Rate Perceived Exertion, Performance Test Parameters and Behaviour During the Different Phases of Menstural Cycle
Brief Title: The Effects of Aerobic Exercise During the Different Phases of Menstural Cycle
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0519
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Menstrual Cycle
Keywords: aerobic exercise; Physical exertion; balance
MeSH Terms: interventions — Patient Education as Topic; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient education (Active Comparator): Patient Education: Providing information on the benefits of physical activity, proper exercise techniques, and self-care strategies. Self-Management Programs: Empowering women to take an active role in managing their health and fitness. Frequency: 3 session/ month, Intensity: Mild to moderate, Type: Walking, Time: 30 to 45mints /sessions
  Interventions: Other: Patient education
- Aerobic exercises (Experimental): Group B will perform the aerobic exercises (such as bicycling, treadmill and running) these exercises. Aerobic exercises performed 30 to 45min/session. Frequency: 3 session /month Intensity: Mild to moderate, Type: treadmill, bicycling, running ,Time: 30 to 45min/month
  Interventions: Other: Aerobics

INTERVENTIONS:
Other: Patient education — The group A will be Education and Self-Management. Patient Education: Providing information on the benefits of physical activity, proper exercise techniques, and self-care strategies.
  Self-Management Programs: Empowering women to take an active role in managing their health and fitness. Frequency: 3 session/ month, Intensity: Mild to moderate, Type: Walking Time: 30 to 45mints /sessions
  Arms: patient education
Other: Aerobics — Treadmill: A manual Treadmill intervention involves moderate-intensity aerobic exercise on a treadmill for 15 minute with the heart rate gradually reaching 75-85% of the maximum. Training frequency was not specified. It significantly reduced menstrual pain intensity 3 session per month. Stationary Bicycling: Start with gentle, low-intensity cycling and gradually increase as comfort allow the duration of exercise 10 mints per month. Running : The running is a low intensity effort of short to moderate duration 10 to 15 mints per mile
  Arms: Aerobic exercises

SUMMARY:
The menstrual cycle is a term to describe the sequence of events that occur in body as it prepares for the possibility of pregnancy each month. The average length of a menstrual cycle is 28 days. However a cycle can range in length from 21 days to about 35 days and still normal. The menstrual cycle is the time from the first day of your menstrual period until the first day of your next menstrual period. Every person's cycle is slightly different, but the process is the same. Menstruation is the monthly shedding of the lining of the uterus. Menstrual blood which is partly blood and partly tissue from the inside of the uterus flows from the uterus through the cervix and out of the body through vagina. Some people experience symptoms of menstruation and others don't. The intensity of these symptoms can also vary. The most common symptom is cramps. The cramping you feel in your pelvic area is your uterus contracting to release its lining. Menstrual cycle have four phases, menses phase (3 to 7 days of your periods), follicular phase (during the 10 to 14 days), ovulation phase (14 day if cycle is 28 days) and luteal phase (15 to 28 days).These will a Randomized control trial conduct on 42 participants. The data will be collected ffrom ladies gym and muscle work gym by using non-probability convenience sampling technique. The age between 18-25 years participants will perform the aerobic exercises during the different phases of menstrual cycle. A sample will be divided into two groups each group have 21 participants. The Group A control group will Education and Self-Management about health and fitness and perform the walk. Group B intervention group will be given the Aerobic exercise (cycling, treadmill and running). The participants assessed with Borg scale for rate perceived exertion, berg balance questionnaire use for performance test parameters and menstrual stress questionnaire use for behaviour. Data will be analyzed by using SPSS version 26.0.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged 18 - 25 years
* Physical active women
* Weight 40 to 60
* Normal BMI ( 18 to 24)

Exclusion Criteria:

* Contraceptive pills
* Perimenupause
* Ammnorehic women
* Pregnant female
* Irregular menstrual cycle
* Non-smokers to minimize confounding cardiovascular effects

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
vertical jump test | baseline and fourth week
  Have each athlete perform between 3 and 5 single, maximal effort jumps, separated by at least 1 minute. Good vertical jump scores vary depending on the type of jump, i.e. counter movement, squat jump, with arms, without arms etc. The following two sets of normative data are both based on vertical jumps being performed with a counter movement and the use of arms.
heart rate | baseline and fourth week
  The point of 6 correlates to a heart rate of 60 beats per minute in a healthy adult, 7 for 70 beats per minute, and so on. The scoring system measures the extreme ranges of exertion on a scale of 6 to 20.

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PHD, Principal Investigator — Riphah International University
Locations (1):
- Sheikh Zayed Hospital,, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bull JR, Rowland SP, Scherwitzl EB, Scherwitzl R, Danielsson KG, Harper J. Real-world menstrual cycle characteristics of more than 600,000 menstrual cycles. NPJ Digit Med. 2019 Aug 27;2:83. doi: 10.1038/s41746-019-0152-7. eCollection 2019. PMID 31482137
- [Background] American Academy of Pediatrics Committee on Adolescence; American College of Obstetricians and Gynecologists Committee on Adolescent Health Care; Diaz A, Laufer MR, Breech LL. Menstruation in girls and adolescents: using the menstrual cycle as a vital sign. Pediatrics. 2006 Nov;118(5):2245-50. doi: 10.1542/peds.2006-2481. PMID 17079600
- [Background] Magyar DM, Boyers SP, Marshall JR, Abraham GE. Regular menstrual cycles and premenstrual molimina as indicators of ovulation. Obstet Gynecol. 1979 Apr;53(4):411-4. No abstract available. PMID 571587